CLINICAL TRIAL: NCT04108169
Title: A Chinese Registry to Evaluate the Association of Surgical Left Atrial Appendage Occlusion vs No Receipt of S-LAAO With Adverse Cardiovascular Events Among Petients Undergoing Coronary Artery Bypass Grafting.
Brief Title: Association Between S-LAAO and Adverse Cardiovascular Events Among Patients Undergoing Coronary Artery Bypass Grafting.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20190926
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Heart Surgery
Keywords: Coronary artery bypass graft; Left Atrial Appendage Occlusion; stroke; prevention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator)
  Interventions: Procedure: Left atrial appendage occlusion surgery
- Sham Comparator (No Intervention)

INTERVENTIONS:
Procedure: Left atrial appendage occlusion surgery — CABG according to indications in the current guidelines on myocardial revascularization including surgical closure of left atrial appendage
  Arms: Active Comparator

SUMMARY:
This is a prospective, single-center, randomized, active controlled, clinical trail to assess the efficacy and safety of surgical closure of left atrial appendage (LAA) in patients undergoing coronary artery bypass graft.

ELIGIBILITY:
Inclusion Criteria:

1. Subject undergoing coronary artery bypass grafting according to clinical indications;
2. Age is more than 18 and less than 80 years old;
3. Male and non pregnancy female;
4. Subject understands study requirements and agrees to sign an informed consent from prior to study procedures.

Exclusion Criteria:

1. Pregnancy female;
2. Participate in other clinical trial in the last 1 month.
3. Subject doesn't agree to sign an informed consent from prior to study procedures.
4. Subject undergoing repeat CABG, concomitant valve or other cardiac surgery.
5. New York Heart Association (NYHA) Class IV heart failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 3 year after discharge (These data is collected during follow-up visit at in-hospital)

SECONDARY OUTCOMES:
Atrial fibrillation | 3 year after discharge (These data is collected during follow-up visit at in-hospital)
Composite of ischemic stroke, thromboembolism and all death | 3 year after discharge (These data is collected during follow-up visit at in-hospital)

CONTACTS AND LOCATIONS:
Overall Officials: Ping Li, PHD, Study Director — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, China